CLINICAL TRIAL: NCT06335992
Title: Activation of Regenerative Pathways by Exercise Training in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Tissue Regeneration in Patients With Chronic Obstructive Pulmonary Disease After an Exercise Intervention.
Acronym: T-Rex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Margareta Emtner, Professor, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2022-00831-01
Record Dates: First submitted 2024-03-07; First posted 2024-03-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Exercise; Regeneration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Experimental): The exercise training protocol to be used in this study:
  Supervised exercise training (aerobic- and muscle strengthening exercise): 2 times a week for 12 weeks.
  * Aerobic exercise with ergometer cycling for 30 min, at moderate intensity (60% Wpeak) individually adjusted to level 4-6 on the Borg category ratio-10 scale.
  * Muscle strengthening exercise will consist of 8-12 strength exercises of the major upper and lower body muscle groups. Each exercise includes three sets with 8-12 repetitions.
  Exercise training at home: once a week for 12 weeks.
  Interventions: Other: Exercise regime

INTERVENTIONS:
Other: Exercise regime — Exercise

SUMMARY:
The main objective of this project is to identify mechanisms for lung regeneration in patients with COPD induced by exercise training. The hypothesis is that adjusted exercise training improves disease outcome in these patients by decrease remodelling processes linked to oxidative stress, inflammatory and/or immunological pathways in the lung. Along the way, the investigator also expect to identify (or validate) biomarkers mirroring systemic processes such as reduced inflammation and ameliorating the epithelial barrier in these patients. These events may additionally act as potential targets for interventions.

Objectives (i) Evaluate biomarkers for regenerative processes, matrix turnover, stem cell activity and inflammatory patterns in lung tissue biopsies, blood- and urine samples correlated to vital lung parameters and physical capacity, before and after attending an exercise-training program.

(ii) Study the effects of exercise training on the pulmonary ventilation/perfusion ratio and quality of life.

(iii) Evaluate the relation between pathophysiology in the lung evaluated by CT scan, and systemic response measured by muscle biopsies and biomarkers in blood/urine.

(iv) Investigate in vitro cell behaviour and remodelling/regenerative processes altered in COPD patients upon exercise training (aim 1).

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is an increasing worldwide health problem characterized by progressive destruction of lung tissue. In the shadow of the pandemic, COPD patients may suffer more severely from COVID-19 with worse prognosis and higher mortality rate. This may be due to common underlying risk factors such as smoking, cardiovascular disease and a sedative life style. To cope with the soaring burden on the health care system posed by the aftermath of the pandemic in the context of chronic diseases such as COPD, the importance of self-responsibility to increase quality of life is emerging. New guidelines from the 2020 GOLD Science Committee Report on COVID-19 and Chronic Obstructive Pulmonary Disease support exercise in the management of COPD and after COVID-19 infection, even during mild COVID-19 symptoms. However, little is known about the molecular alterations induced by exercise training and how to boost the body´s ability to halt disease progression in COPD.

The hypothesize is that adjusted exercise training increases the ability to cope with biological stress, which is increased in COPD due to i.e. chronic inflammation and a history of smoking, and may facilitate restoration of damaged tissue. In this proposal the anticipation is to link the effects of physical exercise to amelioration of vital lung parameters, physical strength including 6 min walk test, and quality of life, by evaluating biomarkers for stem cell activity, regeneration and inflammation in lung tissue biopsies and blood samples. This will also result in the recognition of pathways that are targetable for novel pharmaceuticals that could synergize with the training effect.

ELIGIBILITY:
Inclusion Criteria:

* Forced expiratory volume in one second (FEV1) 85-30 % of predicted post bronchodilator
* Optimal medical treatment according to GOLD and the Swedish National Guidelines
* Absence of other significant diseases that could contribute to physical exercise limitation
* Non-smoking since at least one year
* Free from exacerbations (last 4 weeks)
* BMI = 18- 35

Exclusion Criteria:

* Regular participation in adjusted/specially designed exercise sessions
* Unstable cardiovascular or pulmonary disease
* Smoking
* Any other criteria that at the discretion of the investigator prevent the study subject from participating in an exercise-training program

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function | Baseline, post intervention at 12 wks
  FEV1 (Forced Expiratory volume in one second)

SECONDARY OUTCOMES:
Physical capacity | Baseline, post intervention at 12 wks
  6MWD (six-minute walk distance), longer distance = better health
Inflammation markers | Baseline, post intervention at 12 wks
  Biomarkers (eg. C reactive protein, Interleukin-6)
Level of emphysema | Baseline, post intervention at 12 wks
  HRCT, (high-resolution computed tomography), AiDA (Air space dimension assessment)
Maximal physical capacity ( Wmax) | Baseline, post intervention at 12 wks
  Maximal watt during incremental cardiopulmonary exercise test
COPD Assessment Test (CAT) | Baseline, post intervention at 12 wks
  Health status, Score 1-40, lower score = better health

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Lund University, Lund
  - Uppsala University, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsson C, Elowsson L, Tufvesson E, Cederberg A, Ohrneman H, Falcones B, Karlsson L, Akbarshahi H, Ankerst J, Bjermer L, Palm A, Londahl J, Malinovschi A, Janson C, Emtner M, Westergen-Thorsson G. Activation of regenerative pathways by exercise intervention in subjects with chronic obstructive pulmonary disease - a study protocol. Respir Res. 2025 Dec 12. doi: 10.1186/s12931-025-03443-y. Online ahead of print. PMID 41388411